CLINICAL TRIAL: NCT06310031
Title: Investigation of a Novel, magNetically Levitated VAD for the Treatment of refractOry Left Ventricular heArT failurE
Brief Title: Investigation of the BrioVAD System for the Treatment of Left Ventricular Heart Failure
Acronym: INNOVATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BrioHealth Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-00545
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Heart Failure
Keywords: Heart Failure; Left Ventricular Assist Device; Ventricular Dysfunction; Heart Disease; Cardiovascular Disease; Heart-assist Devices; Left Ventricular Assist System; BrioHealth Solutions
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Failure; Ventricular Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- BrioVAD System (Experimental): BrioVAD® Left Ventricular Assist System (BrioVAD® System) by BrioHealth Solutions, Inc.
  Interventions: Device: BrioVAD System
- HeartMate 3 (Active Comparator): HeartMate 3 System by Abbott
  Interventions: Device: HeartMate 3

INTERVENTIONS:
Device: BrioVAD System — Implantation of the BrioVAD System to evaluate the safety and efficacy of the BrioVAD System by demonstrating non-inferiority to the HeartMate 3 LVAS when used for the treatment of advanced, refractory, left ventricular heart failure.
  Arms: BrioVAD System
Device: HeartMate 3 — Implantation of the commercially approved HeartMate 3 LVAS, which is the standard treatment for advanced heart failure.
  Arms: HeartMate 3

SUMMARY:
The goal of this study is to evaluate the safety and efficacy of the BrioVAD System by demonstrating non-inferiority to the HeartMate 3 Left Ventricular Assist System when used for the treatment of advanced, refractory, left ventricular heart failure.

DETAILED DESCRIPTION:
The INNOVATE Trial is a prospective, non-blinded, randomized, controlled, multi-center, non-inferiority study to evaluate the safety and efficacy of the BrioVAD System by demonstrating non-inferiority to the HeartMate 3™ (HM3) LVAS (Abbott) when used for the treatment of advanced, refractory left ventricular heart failure. It is the first clinical study to compare two left ventricular assist devices (LVAD) that belong to the same category of fully magnetically levitated LVAD.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years of age.
2. Patient has received institutional approval for LVAD implantation.
3. Patient has a body surface area (BSA) ≥ 1.2 m2.
4. Patient is classified as NYHA Class IV with advanced heart failure refractory to advanced heart failure management or NYHA Class III with dyspnea upon mild physical activity.
5. Patient has a left ventricular ejection fraction (LVEF) ≤ 25% or LVEF < 30% on inotropes or temporary MCS.
6. Patient is inotrope dependent, OR has a cardiac index (CI) ≤ 2.2 liters/min/m2, while not on inotropes, and also meets one of the following criteria:

   1. Is on optimal medical management (OMM), based on current heart failure practice guidelines for at least 45 out of the last 60 days and is failing to respond or is not able to tolerate OMM; or
   2. Has advanced heart failure for at least 14 days and is dependent on an intra-aortic balloon pump (IABP) or temporary mechanical circulatory support device (MCSD) for at least seven days.
7. Patient has provided voluntary and informed consent.
8. Females of childbearing age agree to use adequate contraception and have a negative pregnancy test.

Exclusion Criteria:

1. Patient's heart failure etiology is related to restrictive or constrictive physiology (e.g., nondilated hypertrophic cardiomyopathy, cardiac amyloidosis/senile or other infiltrative disease), complex congenital heart disease (e.g., transposition of the great vessels), uncorrected thyroid disease, and/or pericardial disease.
2. Patient had a myocardial infarction within seven days of study enrollment.
3. Patient had cardiothoracic surgery within 30 days of implant with the exception of a procedure to implant temporary MCS: Impella 5.5, Impella CP or TandemHeart.
4. Patient has physiological conditions or comorbidities which pose high surgical risk or obstacles as determined by the Investigator.
5. Patient has contraindications to warfarin anticoagulation.
6. Patient has known hypo- or hypercoagulable state [e.g., disseminated intravascular coagulation (DIC)], or has a positive heparin-induced thrombocytopenia (HIT) assay and positive serotonin release assay or requires use of a non-heparin alternative anticoagulation strategy for cardiopulmonary bypass in the judgement of the Investigator.
7. Patient is on durable MCS (e.g., LVAD or RVAD).
8. Planned need for durable or temporary RVAD support concomitant with LVAD implant.
9. Patient is on any form of pre-implant temporary MCS other than isolated LVAD support with an intra-aortic balloon pump, Impella 5.5, Impella CP, or TandemHeart.
10. Patient is on any form of pre-implant temporary MCS and has a serum lactate dehydrogenase greater than 2.5 times the upper limits of normal or plasma free hemoglobin > 40 g/dL.
11. Patient has a history of organ transplantation.
12. Patient has a mechanical aortic valve that may not be converted to a bioprosthetic valve at the time of VAD implant.
13. Patient has a platelet count < 50 k/μl.
14. Patient has a history of confirmed untreated abdominal aortic aneurysm (AAA) > 5 cm in diameter.
15. Patient has moderate or severe aortic insufficiency that will not be corrected during the VAD implant procedure.
16. Patient has an uncontrolled systemic infection.
17. Patient has a positive COVID 19 test within 21 days of study enrollment and at least one high risk feature including need for supplemental oxygen or ferritin >1000 ug/L.
18. Patient has severe end-organ dysfunction as evidenced by one or more of the following criteria:

    1. Total bilirubin > 3.0 mg/dL or cirrhosis confirmed by liver imaging or hemodynamic assessment with or without biopsy confirmation.
    2. International normalized ratio (INR) ≥ 2.0 or PTT > 2.5 times control that is not related to anticoagulation therapy.
    3. Glomerular filtration rate (GFR) < 30 mL/ min/1.73 m2 or need for renal replacement therapy.
    4. Severe pulmonary arterial hypertension with a pulmonary vascular resistance (PVR) ≥ 8 Wood units that is not acutely reversible with pharmacologic intervention.
    5. Severe chronic obstructive pulmonary disease (COPD) or restrictive lung disease requiring home oxygen or an FEV1/FVC < 0.7 and FEV1 < 40% predicted.
    6. Mechanical ventilation for more than three days present at the time of study enrollment.
    7. Documented history of pulmonary embolism or pulmonary infarct within 60 days of study enrollment.
    8. History of stroke within 90 days of study enrollment or history of stroke with a mRS ≥ 3 at the time of study enrollment.
    9. Symptomatic cerebrovascular disease and/or uncorrected carotid stenosis > 80%.
    10. Significant peripheral vascular disease (PVD) accompanied by pain at rest or extremity ulceration.
    11. Pre-albumin < 15 mg/dL and/or albumin < 2.5 g/dL.
19. Patient has a non-cardiac comorbidity or illness that would limit survival to less than two years.
20. Patient has a psychiatric disease or disorder, or irreversible cognitive dysfunction, and/or insufficient social support or a history of non-adherence with medical instructions that is likely to impair study compliance.
21. Patient is participating in an interventional clinical trial that may impact or confound the results of the INNOVATE Trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Short-Term Indication Primary Endpoint | 6 months
  Composite of survival to transplant, recovery or 6 months of LVAD support free of debilitating stroke [modified Rankin Scale (mRS) > 3], or reoperation to replace the pump
Long-Term Indication Primary Endpoint | 24 months
  Composite of survival to transplant, recovery or 24 months of LVAD support free of debilitating stroke (mRS > 3), or reoperation to replace the pump.

SECONDARY OUTCOMES:
Powered Secondary Endpoint | 24 months
  Total number of nights in hospital, skilled nursing facility, or inpatient rehabilitation, inclusive of index hospitalization, through 24 months post VAD implant, heart transplantation, VAD explant or decommission, study withdrawal, or death, whichever occurs first.
Short-Term Indication Secondary Endpoint | 6 months
  Evaluation of the short-term safety using INTERMACS adverse event (AE) terms and definitions through 6 months post VAD implant, heart transplantation, VAD explant or decommission, study withdrawal, or death, whichever occurs first. Incidences of all AEs and the event rate per patient year of support through 6 months will be reported. Differences in the event rates between the Study Arm and the Concurrent Control Arm will be analyzed. Serious adverse events (SAEs) will be analyzed in a similar manner.
Long-Term Indication Secondary Endpoint | 24 months
  Evaluation of the long-term safety using INTERMACS AE terms and definitions through 24 months post VAD implant, heart transplantation, VAD explant or decommission, study withdrawal, or death, whichever occurs first. Incidences of all AEs and the event rate per patient year of support through 24 months will be reported. Differences in the event rates between the Study Arm and the Concurrent Control Arm will be analyzed. SAEs will be analyzed in a similar manner

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Baptist Health Medical Center-Little Rock, Little Rock, Arkansas
  - UF Health Shands Hospital, Gainsville, Florida
  - Advent Health, Orlando, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Advocate Christ Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Ascension St. Vincent Hospital - Indianapolis, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health, Detriot, Michigan
  - Corewell Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - NYU Langone Health, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - The Christ Hospital - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Baptist - Memphis (Stern), Memphis, Tennessee
  - Baylor University Medical Center, part of Baylor Scott & White Health, Dallas, Texas
  - Baylor Scott & White Medical Center - Plano, Plano, Texas
  - University of Utah, Salt Lake City, Utah
  - Inova Fairfax Medical Campus, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
Protocol and data is company confidential.